CLINICAL TRIAL: NCT07145138
Title: University of Illinois Chicago (UIC) Multi-Ethnic Dilated Cardiomyopathy (DCM) Registry
Brief Title: UIC Multi-Ethnic DCM Registry
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, David Tofovic, Assistant Professor, University of Illinois at Chicago
Other Study IDs: STUDY2023-0255
Record Dates: First submitted 2025-04-08; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Dilated Cardiomyopathy (DCM)
Keywords: Dilated Cardiomyopathy; Heart Failure; Genomics; Social Determinants of Health; Variant
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dilated Cardiomyopathy
- Control

SUMMARY:
Dilated cardiomyopathy (DCM), a condition where the heart loses its ability to pump blood throughout the body, is a common cause of death in the United States (US). It affects minorities more frequently and appears to causes greater harm than Whites. However, almost all research related to DCM has been performed in Whites, where up to half of cases run in the family. Several genes have been identified that cause the disease, but we are unsure if these same genes are also responsible for DCM in African Americans or Hispanic/Latino patients. The impact of various medical, social, and financial stressors on the severity of the disease in ethnic minorities also remains unclear. The investigators believe that certain genes are more common in different racial and ethnic groups and the greater medical, social, and financial burden faced by minorities in the US leads to more harm from DCM in these groups. The overall goal of the project is to test whether ethnic minority patients carrying genes that cause DCM experience more adverse effects in part because of various medical, social, and financial burdens. The investigators will first establish the UIC Multi-ethnic DCM Biorepository to look for how often certain genes are found across different race-ethnicity and then ask the question if these genes impact the severity of DCM. Finally, the investigators will study how a person's environment can alter the course of their disease. Through this, the investigators hope and strive to ensure equal and adequate heart care for individuals regardless of their race-ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age and be admitted to or seen at a UIH site.
* Subjects must be willing and able to give written, informed consent

Exclusion Criteria:

* Adults who are unable to provide consent
* Women who are pregnant at the baseline visit,
* Prisoners
* Individuals who are not yet adults (infants, children, teenagers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Only nonpregnant and noninstitutionalized adults will be considered for study enrollment. Two separate groups of patients will be eligible for study enrollment, those without a history of DCM (i.e. controls) and those with an identified history of DCM (i.e. cases). Clinic lists, inpatient team lists, and echocardiography lab lists will be surveyed daily by study coordinators to identify potential enrollees. Subjects will be approached for potential enrollment during outpatient visits to either the Family Medicine clinics, Internal Medicine clinics, or one of the four outpatient Cardiology Clinic or during inpatient stay at University of Illinois Hospital. Patients will be categorized as having DCM based on clinically report history or a transthoracic echocardiography (TTE) or cardiac magnetic resonance imaging (CMRI) showing LVEF <50% and LV end-diastolic diameter (LVEDD) ≥95th percentile, meeting criteria for DCM.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2038-12-31 (Estimated)

PRIMARY OUTCOMES:
Likely Pathogenic/Pathogenic Variants | Baseline
  Utilizing genomic sequencing, the investigators will obtain blood samples at baseline for study participants and identify utilizing genomic sequencing the prevalence of likely pathogenic/pathogenic (LP/P) variants in dilated cardiomyopathy patients across race-ethnicity.

SECONDARY OUTCOMES:
Severity of Disease Symptoms: Minnesota Living with Heart Failure Questionnaire (MLHFQ) Score | Participants with heart failure or who develop heart failure will complete the digital MLHFQ assessments at 12 months, 24 months, and 60 months after initial enrollment or new heart failure diagnosis.
  Minnesota Living with Heart Failure Questionnaire (MLHFQ) Score will be administered to study participants with heart failure at set time points to access symptom burden. Score is based on a range of 0 to 105, with lower scores corresponding to lower symptom burden.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Hospital & Health Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Access to trial IPD can be requested by qualified researchers engaging in independent scientific research within the University of Illinois Chicago (UIC) and outside (non-UIC) interrogators in the future for research purposes only. These requests will be subject to IRB approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA) at UIC and any outside institution.